CLINICAL TRIAL: NCT02623153
Title: Phase 2 Study of Comparison Between XELOX (Capecitabine and Oxaliplatin) and Docetaxel, Oxaliplatin and S1 Regimen as Neoadjuvant Chemotherapy for Patients With Locally Advanced Gastric Cancer
Brief Title: Comparison Between XELOX and S1, Oxaliplatin and Docetaxel as Neoadjuvant Chemotherapy for Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianshu Liu (Other)
Responsible Party: Sponsor-Investigator, Tianshu Liu, Chairman of the department of oncology, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zswy003
Record Dates: First submitted 2015-11-28; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine; S 1 (combination); Tegafur; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- capecitabine and oxaliplatin (Active Comparator): capecitabine of 1000 mg/m2, orally administered twice a day on days 1-14 and oxaliplatin at 130 mg/m2on day 1, as intravenous 2 h infusion
  Interventions: Drug: Oxaliplatin; Drug: capecitabine
- S1, oxaliplatin and docetaxel (Experimental): S1 of 40 mg/m2, orally administered twice a day on days 1-14,oxaliplatin 130 mg/m2 and docetaxel 40 mg/m2on day 1 as intravenous
  Interventions: Drug: Oxaliplatin; Drug: S1; Drug: Docetaxel

INTERVENTIONS:
Drug: Oxaliplatin — oxaliplatin 130 mg/m2
  Other Names: Eloxatin
Drug: capecitabine — capecitabine of 1000 mg/m2
  Other Names: Xeloda
  Arms: capecitabine and oxaliplatin
Drug: S1 — S1 of 40 mg/m2
  Other Names: tegafur
  Arms: S1, oxaliplatin and docetaxel
Drug: Docetaxel — docetaxel 40 mg/m2
  Other Names: Taxotere
  Arms: S1, oxaliplatin and docetaxel

SUMMARY:
The choice of neoadjuvant chemotherapy regimen for locally advanced gastric cancer is controversial. The aim of this study was to compare the short- and long-term outcomes of XELOX regimen with Docetaxel, S1 and oxaliplatin regimen as neoadjuvant chemotherapy regimen for locally advanced gastric cancer. The objective of this study is to determine what kind of neoadjuvant chemotherapy strategy can make subsequent radical surgery feasible and improve overall survival in patients with locally advanced gastric cancer.

DETAILED DESCRIPTION:
Patient selection

Patients with unresectable, histologically confirmed gastric adenocarcinoma with no distant metastases were eligible for the study. No-resectability was judged for technical reasons by a local multidisciplinary team, according to one of the following criteria:

1. radical resection was unable after laparotomy or laparoscopic exploration.
2. tumour invades adjacent structures such as the pancreas, liver, diaphragm, adrenal gland or transversa colon (T4b).
3. Para-aortic (LN)lymph node metastasis ≥1.0 cm between the upper margin of the celiac artery and the upper border of the inferior mesenteric artery(stations no. 16a2/16b1), and/or bulky lymph nodes (≥3 cm×1 or≥1.5 cm×2) along the celiac, splenic, common or proper hepatic arteries, or the superior mesenteric vein;

All the patients received endoscopic examination, contrast CT scan for abdomen and pelvic, chest X-ray, as well as physical examination.

The exclusion criteria included: (1)peritoneal metastasis confirmed by CT scan; (2) lung metastasis, liver metastasis, pleural effusion, and/or other distant metastasis; (3) serious uncontrolled comorbid conditions; (4)any local intervention after initial diagnosis, such as surgical procedures, radiotherapy or trans-artery chemo-embolization;(5) patients who could not comprehend or comply with the study were also ineligible.

A multidisciplinary evaluation was required before any patient's participation in this study. All patients signed an approved written informed consent. The protocol of this trial was approved by the institutional review board of Zhongshan Hospital, Fudan University.

Preoperative chemotherapy All the patients received chemotherapy after diagnosis. Since no definite regimens are instructed by the guideline, physicians prescribed XELOX regimen (capecitabine of 1000 mg/m2, orally administered twice a day on days 1-14 and oxaliplatin at 130 mg/m2on day 1, as intravenous 2 h infusion) or S1 of 40mg/m2, orally administered twice a day on days 1-14,oxaliplatin at 130 mg/m2 and docetaxel 40 mg/m2on day 1 as intravenous according to the clinician's preference. Chemotherapy was repeated every three weeks.

Tumor response and toxicity criteria After every two cycles (6 weeks), an abdominal and pelvic CT scan was performed to evaluate the tumor response.Treatment was planned for four cycles after which tumors were assessed for the respectability by a multidisciplinary team using CT scan. Resection was intended to be done within 4-6 weeks of the last treatment cycle. Patients with unresectable tumors continued treatment until tumor response progression, and were assessed for respectability every two cycles for a maximum duration of eight cycles. Following resection, patients were continued on treatment for four cycles. . Patients with progressive disease or unacceptable toxicity were treated at the discretion of the investigators.Response to the treatment was evaluated according to response evaluation criteria in solid tumor (RECIST) 1.1. The adverse events were assessed according to the Common Toxicity Criteria of the National Cancer Institute (NCI-CTC) 3.0.

Surgical procedure The type of surgery performed depended on the location and extent of the primary cancer. The tumor was resected along with a gastric margin of ≥5 cm when feasible. For a distal tumor, a subtotal gastrectomy was considered, and total gastrectomy was performed for proximal cancers. An attempt was made to perform an extended LN(lympho node) resection (D2) in any patient who was qualified to go under-radical surgery. The surgical specimens were pathologically evaluated as grade0 when degeneration and/or necrosis were absent with in the tumor, grade 1a when these areas accounted for less than one-third of the tumor, grade 1b when these areas accounted for more than one-third and less than two-thirds of the tumor, grade 2a when these areas accounted for more than two-thirds of the tumor, although tumor tissue apparently remained, grade 2b when only minimal tumor cells remained, and grade 3 when no residual tumor was detected.Patients with grade 1b, 2a, 2b, or 3 tumors were classified as responders, while pathologic complete response (pCR) was defined as grade 3.

Postoperative treatment After R0 resection, adjuvant chemotherapy with the original regimen was initiated within 42 days of surgery, and eight cycles were administered during perioperative period. Patients who could not undergo a radical operation received palliative chemotherapy until evidence of disease progression appeared. All enrolled patients were followed up regularly. Physical and blood examinations were conducted every 3 months for the first 3 years and every 6 months thereafter. An abdominal CT scan was performed every 6 months for the first 3 years, and every year thereafter. Chest CT scan and upper gastrointestinal endoscopy were conducted every year.

Statistical analysis The primary study endpoint was the response rate, and secondary endpoints included R0 resection rate, progression-free survival (PFS), overall survival (OS) and toxicity. PFS was measured from the date of initial treatment to the first objective documentation of disease progression, palliative surgery or relapse. OS was measured from the start of the treatment to the date of the last follow-up or death. All patients were followed up every three months.

Patient baseline characteristics and disease factors were summarized using descriptive statistics. The categorical parameters were compared using two-sided Pearson's test or Fisher's exact test, as appropriate.The PFS and OS were generated by the Kaplan-Meier method and were compared by means of the log-rank test. Software(version 16.0; Chicago, IL) was used for statistical analyses. A P<0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with unresectable, histologically confirmed gastric adenocarcinoma with no distant metastases were eligible for the study.

Exclusion Criteria:

* peritoneal metastasis confirmed by CT scan
* lung metastasis, liver metastasis, pleural effusion, and/or other distant metastasis
* serious uncontrolled co-morbid conditions
* lacking of measurable target lesion
* any local intervention after initial diagnosis, such as surgical procedures, radiotherapy or trans-artery chemo-embolization
* patients who could not comprehend or comply with the study were also ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
response rate | through study completion, an average of 24 weeks

SECONDARY OUTCOMES:
R0 resection rate | through study completion, an average of 24 weeks
progression-free survival | through study completion, an average of 1 year
overall survival | through study completion, an average of 2 year
adverse events | through study completion, an average of 1 year